CLINICAL TRIAL: NCT04291924
Title: Validity and Reliability of a Low-cost Chair Dynamometer
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Spinal Cord Injury Centre of Western Denmark (Other)
Collaborators: University of Aarhus (Other)
Responsible Party: Principal Investigator, Søren Krogh Jensen, Principal Investigator, Spinal Cord Injury Centre of Western Denmark
Other Study IDs: VALREL DYNAMOMETER
Record Dates: First submitted 2020-02-27; First posted 2020-03-02 (Actual); Last update posted 2020-10-27 (Actual); Status verified 2020-10

CONDITIONS: Spinal Cord Injuries
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Ablebodied individuals
  Interventions: Diagnostic Test: Dynamometry
- Spinal Cord Injured Individuals
  Interventions: Diagnostic Test: Dynamometry

INTERVENTIONS:
Diagnostic Test: Dynamometry — A test for maximal muscle strength and explosive power in the lower limbs

SUMMARY:
In part 1 of the study, fourteen able-bodied individuals will undergo maximal, voluntary contraction (MVC) test of the lower limbs in two dynamometers. One being a low-cost dynamometer (S2P-CD), and the other being a gold standard dynamometer (HUMAC). Thereby the investigators will be able to assess the validity of the S2P-CD.

In part 2 of the study, eighteen persons with spinal cord injury will undergo MVC twice in the S2P-CD. Thereby the investigators will be able to assess the reliability of the measurements of the S2P-CD.

DETAILED DESCRIPTION:
In part 1 of the study, fourteen able-bodied individuals will undergo maximal, voluntary contraction (MVC) test of the lower limbs in two dynamometers. One being a low-cost dynamometer (S2P-CD), and the other being a gold standard dynamometer (HUMAC). The tests will be carried out with 72-96 hours between them. Thereby the investigators will be able to assess the validity of the S2P-CD.

In part 2 of the study, eighteen persons with spinal cord injury will undergo MVC twice in the S2P-CD. Participants will be recruited through the Spinal Cord Injury Centre of Western Denmark (SCIWDK). The test will be carried out with 30min between them. Thereby the investigators will be able to assess the reliability of the measurements of the S2P-CD.

ELIGIBILITY:
Ablebodied individuals:

Inclusion Criteria:

* Age >18 y

Exclusion Criteria:

* Orthopedic or other injuries that may limit maximal muscle strength

Spinal cord injured individuals:

Inclusion Criteria:

* Age > 18 y
* Congenital or acquired spinal cord injury with some degree of preserved muscle function in the lower limbs

Exclusion Criteria:

* Orthopedic or other injuries that may limit maximal muscle strength
* Significant competing diseases
* Severe osteoperosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Ablebodied, healthy volunteers
  Spinal cord injured individuals admitted at SCIWDK
Sampling Method: Probability Sample
Enrollment: 32 (Estimated)
Dates: Start 2020-11-15 (Estimated); Primary Completion 2021-02-01 (Estimated); Study Completion 2021-04-01 (Estimated)

PRIMARY OUTCOMES:
Maximal voluntary contraction | 15min
  Maximal muscle strength

SECONDARY OUTCOMES:
Rate of force development | 15min
  Explosive muscle strength

CONTACTS AND LOCATIONS:
Overall Officials: Søren K Jensen, MSc, Principal Investigator — Spinal Cord Injury Centre of Western Denmark
Locations (1):
- Spinal Cord Injury Centre of Western Denmark, Viborg, Denmark

IPD SHARING:
Plan to Share IPD: No